CLINICAL TRIAL: NCT05920603
Title: Iodine Status of the Indigenous Peoples (Karen) Living in Laiwo Subdistrict, Sangkhlaburi District, Kanchanaburi Province, Thailand
Brief Title: Iodine Status of the Indigenous Peoples (Karen) Living in Thailand
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Iodine Global Network (Unknown); ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: MU-CIRB 2022/178.3006
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Iodine Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- School-aged children (6-12 years old) and women of reproductive age (15-49 years old): 300 healthy school-aged children (6-12 years old), and 300 healthy reproductive-aged women, aged (15-49 years old)

SUMMARY:
In describing the iodine status involving health conditions of the minority groups, this observational study aims to learn about the iodine status of the Indigenous Peoples (Karen) in a subdistrict in western Thailand. The Participants will be collected their urine to determine urinary iodine concentrations At the same time, their household salt will be also collected to determine iodine content.

DETAILED DESCRIPTION:
Iodine deficiency (ID) is a global public health problem, and it is estimated that almost 240 million school-aged children (SAC) worldwide have an insufficient iodine intake. Currently, severe ID is uncommon, but mild-to-moderate ID is still widespread on a global level, especially in the Asia region. Iodine deficiency causes multiple adverse effects on growth and development in all age groups. Salt iodization is recommended as the most cost-effective way of delivering iodine to the target population to combat iodine deficiency. In addition, the cyclic monitoring of urinary iodine concentration (UIC) in vulnerable groups is recommended by the World Health Organization (WHO).

However, some minority communities such as indigenous peoples living in remote rural areas are not included in IDD surveillance programs. Indigenous peoples in many developing countries, including Thailand, are largely ignored in development efforts, as they are disadvantaged minority groups in those societies. These indigenous peoples may therefore be at risk of many adverse health and nutrition consequences, resulting in their quality of life. In order to promote nutrition and health, and to ensure adequate iodine intake among indigenous peoples in Thailand, it is essential to understand the urinary iodine concentration of the populations and the iodine content in their household salt. The results from this study could then be considered and potentially strengthen the Universal Salt Iodization (USI) program in Thailand, to reach indigenous peoples in border areas.

This study will conduct in Karen communities in Laiwo Subdistrict, Sangkhlaburi District, Kanchanaburi Province, Thailand. The participants will be divided into 2 groups, school-aged children, males and females (6-12 years), and women of reproductive age (15-49 years). The Participants will be collected their urine to determine urinary iodine concentrations At the same time, their household salt will be also collected to determine iodine content.

ELIGIBILITY:
Inclusion Criteria:

* Karen ethnic population living in Laiwo Subdistrict, Sangkhlaburi District, Kanchanaburi Province, Thailand
* Healthy school-aged children, male and female, aged 6 -12 years old (n=300)
* Healthy reproductive-aged women, aged 15 - 49 years old (n=300)
* Can follow the steps of this study

Exclusion Criteria:

* NO

Ages: 6 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — * school-aged children (6-12 years) group recruited both male and female
  * women of reproductive age (15-49 years) group recruited only female
Study Population: The participants are the Karen ethnic population living in Laiwo Subdistrict, Sangkhlaburi District, Kanchanaburi Province, Thailand. It is located in the Thungyai Naresuan National Wildlife Sanctuary some 336 km northwest of Bangkok adjacent to the Myanmar border, and about 12 km east of Sangkhlaburi municipality. The participants are divided into 2 groups, including school-aged children, males and females (6-12 years old), and women of reproductive age (15-49 years old).
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration | 1 day
  A spot urine samples will be collected from each participant at school or their home or a nearby village health promoting hospital. The urine samples will be transported on ice to the Institute of Nutrition of Mahidol University (INMU), divided into aliquots, and stored at -20ºC until analysis. At INMU, the iodine concentration in urine will be measured using the Pino modification of the Sandell-Kolthoff reaction.

SECONDARY OUTCOMES:
Iodine content in salt | 1 day
  The participants will be requested to bring 2 tablespoons of the salt which is commonly consumed in their household, in a tightly sealed plastic bag given by study team. The salt samples will be transported to the Institute of Nutrition of Mahidol University (INMU), and stored under dry conditions until analysis. At INMU, the iodine content in salt will be measured using iodometric titration technique.

CONTACTS AND LOCATIONS:
Overall Officials: Sueppong Gowachirapant, Ph.D., Principal Investigator — Mahidol University
Locations (1):
- Sanaephong, Kongmongta, and Koh Sadueng Villages, Kanchanaburi, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmermann MB, Jooste PL, Pandav CS. Iodine-deficiency disorders. Lancet. 2008 Oct 4;372(9645):1251-62. doi: 10.1016/S0140-6736(08)61005-3. PMID 18676011
- [Background] Andersson M, Karumbunathan V, Zimmermann MB. Global iodine status in 2011 and trends over the past decade. J Nutr. 2012 Apr;142(4):744-50. doi: 10.3945/jn.111.149393. Epub 2012 Feb 29. PMID 22378324
- [Background] Zimmermann MB, Andersson M. GLOBAL ENDOCRINOLOGY: Global perspectives in endocrinology: coverage of iodized salt programs and iodine status in 2020. Eur J Endocrinol. 2021 Jun 10;185(1):R13-R21. doi: 10.1530/EJE-21-0171. PMID 33989173
- [Background] Pino S, Fang SL, Braverman LE. Ammonium persulfate: a safe alternative oxidizing reagent for measuring urinary iodine. Clin Chem. 1996 Feb;42(2):239-43. PMID 8595717
- See also: World Health Organization. Assessment of iodine deficiency disorders and monitoring their elimination. Geneva: World Health Organization, 2007. — http://apps.who.int/iris/bitstream/handle/10665/43781/9789241595827_eng.pdf?sequence=1&isAllowed=y